CLINICAL TRIAL: NCT03731351
Title: Mild Acute Ischemic Stroke With Large Vessel Occlusion (MIST WAVE)
Brief Title: Mild Acute Ischemic Stroke With Large Vessel Occlusion (MISTWAVE)
Acronym: MISTWAVE
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Gabor Toth, MD, Vascular and Interventional Neurologist, The Cleveland Clinic
Other Study IDs: 16-685
Record Dates: First submitted 2018-09-04; First posted 2018-11-06 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Large Vessel Occlusion; mechanical thrombectomy; acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — Acute Ischemic Stroke patient with Large Vessel Occlusion and NIHSS less than or equal to 5 will have a standard of care mechanical thrombectomy. Mechanical thrombectomy is a treatment for stroke that removes clots that block large blood vessels. Some patients may be candidates for this procedure using an angiogram or a catheterization and a device that grabs clots and removes them, to reestablish blood flow to the brain.

SUMMARY:
Stroke remains the leading cause of disability in the United States. An estimated 40-50% of all ischemic strokes are caused by large-vessel occlusion of a major cerebral artery (LVO). However, in some cases, the occlusion results in mild symptoms, at least initially, and these patients frequently do not receive any treatment. These strokes, however, may result in unfavorable long-term outcomes despite relatively benign initial course. Recent large randomized studies in patients with severe stroke symptoms and associated LVO showed efficacy and safety of endovascular mechanical thrombectomy, but patients with mild symptoms were not specifically addressed.

Based on the investigators' own data and limited evidence in the literature, the investigators propose that early mechanical thrombectomy in patients with LVO associated with mild stroke symptoms (defined as NIHSS ≤ 5) is safe, and results in favorable long-term patient outcomes.

The objective of this prospective pilot study is to assess the safety and outcomes of mechanical thrombectomy in patients presenting with acute ischemic stroke due to a large vessel occlusion in the anterior or posterior circulation under 24 hours with mild symptoms (NIHSS ≤ 5).

DETAILED DESCRIPTION:
Patients who present with mild stroke symptoms (mAIS), and are also found to have an intracranial large vessel occlusion (LVO) pose an exceptionally difficult therapeutic dilemma. The need for any acute treatment is often debated since these patients "only" have mild deficits, and any therapy has associated risks. However, it has been shown that acute ischemic stroke (AIS) can lead to considerable morbidity and mortality even in patients presenting with mild symptoms (mAIS) in the presence of LVO. Despite reports that such patients have less favorable outcomes, these patients are often excluded from acute stroke therapy. Recent studies demonstrated that, despite mild and rapidly improving symptoms, many patients end up with unfavorable outcome. While the most recent AHA/ASA guidelines no longer recommend excluding patients with milder improving symptoms from intravenous tissue plasminogen activator administration, the role of endovascular intervention has not been clarified for these patients.

Prior data has shown high morbidity and mortality in mAIS patients (without specified large vessel status), who did not receive IV tPA, demonstrating that as high as 32% of patients was dependent during discharge or died in one study. A common reason for foregoing treatment in this patient group was that mild symptoms or rapid improvement were a contraindication to IV-tPA administration according to previous ASA/AHA guidelines. Higher morbidity was specifically noted in patients with concurrent large vessel occlusion as a cause of the symptom in another study. Mokin et al showed that for LVO patients excluded from thrombolysis, only 2/3rd could walk independently at discharge.

When assessing predictors of poor outcome, LVO seems to correlate with poor outcome despite mild symptoms. Nedeltchev et al published a study with 162 patients with either mild stroke symptoms (NIHSS of 3 or less) or rapidly improving symptoms (NIHSS improvement of 4 points or more), in which 25% of the patients had an unfavorable outcome. NIHSS of 10 or more and proximal vessel occlusion were independent predictors of poor outcome. LVO in patients with rapidly improving /mild symptoms conferred an 18-fold increased risk of early neurological deficit with infarct expansion. Patients with LVO were also more likely to have increased modified ranking scale (mRS), and LVO was an independent predictor of decline in functional status and a borderline significant predictor of poor outcome when adjusting for age, gender and presenting NIHSS.

NIH Stroke Scale Score Threshold The ideal NIHSS cutoff value for "mild" stroke remains unclear, and varies across studies. The investigators specifically chose the NIHSS 5 cut-off value for the cohort after careful consideration of the results of several earlier reports, which were available at the initiation of our research project. These studies, albeit with limited sensitivity and specificity, have concluded that an NIHSS cut-off of 7-10 and higher might be a reliable predictor of LVO. Since the investigators were trying to capture a controversial stroke population that was unlikely to have LVO because of mild symptoms, the investigators decided to include patients with NIHSS 5 or less.

Currently approved treatment and limitations At present, the American Heart Association and American Stroke Association guidelines recommend that eligible ischemic strokes be treated with IV tissue plasminogen activator (tPA) and/or mechanical thrombectomy. Severity of the stroke is based on the National institute of health stroke scale (NIHSS), and the guidelines do not specify any thrombolysis treatment for mild strokes.

Mechanical thrombectomy using stent retrievers for LVO stroke has become the standard of care; however, current guidelines exclude patients with mild or improving symptoms. These recommendations were made based on the 2015 randomized control trials, most of which did not include patients with NIHSS <6.

Despite the MR-CLEAN trial's inclusion of patients with NIHSS as low as 2, which showed efficacy of IAT for LVO, it is unclear what proportion of successfully treated patients were actually in the mAIS category. The PRISMS study investigated the efficacy IV-tPA in mAIS patients, although establishment of large vessel status was not specifically required (NCT02072226). The TEMPO -1 trial showed safety and feasibility of tenecteplase in patients with LVO and mAIS, and the TEMPO - 2 trial (NCT02398656) comparing tenecteplase to standard therapy is currently ongoing.

The recently completed DAWN trial is an international multi-center randomized trial study of patients with acute ischemic anterior stroke due to large vessel occlusions between 6 -24 hours of stroke with endovascular therapy. The results from 206 patients enrolled in the trial demonstrated treatment with use of stentriver significantly decreased post-stroke disability and improved functional independence at 90 days when compared to medical management alone (48.6% vs 13.1%, p<0.001), a relative reduction in disability of 73% percent. The study showed that one in 2.8 patients treated with the stentriever within 24 hours of a stroke is saved from severe disability. Another large trial, the Diffusion and Perfusion Imaging Evaluation for Understanding Stroke Evolution 3 (DEFUSE 3), was halted after the DAWN trial results were presented. This study enrolled patients with large vessel occlusion presenting within 6 and 16 hours of stroke onset based on advanced imaging criteria. Patients who underwent endovascular therapy had 2.77 times greater odds of regaining functional independence at 90 days, versus medical management alone (45% vs 17%, p<0.001), showing benefit for the endovascular group.

Acute vertebrobasilar occlusion The efficacy of mechanical thrombectomy in the anterior circulation raised the question of its potential applicability in the posterior circulation. Acute basilar occlusion accounts for approximately 1% of all acute ischemic strokes, and is disproportionately associated with a mortality rate of approximately 70%. Given these statistics, procedural risks in acute basilar occlusion syndromes have long been regarded much lower than the risk of unfavorable outcome without intervention. Therefore these patients have largely been omitted from clinical trials resulting in a paucity of clinical evidence, in contrast with anterior circulation strokes. Patients with mild-to-moderate posterior circulation AIS pose a unique challenge, as retrospective data correlate the patients' clinical outcome with severity at presentation, giving them up to 67% chance of achieving a favorable outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 85.
2. Clinical signs consistent with acute ischemic stroke.
3. No prestroke functional dependence (prestroke Modified Rankin Score ≤ 1).
4. NIHSS <6 at the time of enrollment.
5. Consent obtained within 24 hours from last known well.
6. Thrombolysis in Cerebral Infarction (TICI) 0-1 flow in

   1. The M1 or M2 segment of the MCA, or carotid terminus confirmed by CT or MR angiography; or
   2. The basilar artery.
7. Subject can be treated within 1 hours (60 minutes) from pre-procedure CT or MRI to groin puncture.
8. CT or MRI-DWI ASPECT Score of > 6 in the anterior circulation, or posterior circulation ASPECT Score (pc-ASPECTS) of > 7.36
9. Subject is willing to conduct protocol-required follow-up visits.
10. Subject or subject's legally authorized representative has signed and dated an Informed Consent Form.

NB: Patient can be enrolled regardless of whether the patient received IV t-PA. However, the decision for administration of IV t-PA must be made before enrolling into the study.

Exclusion Criteria:

1. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
2. Known serious sensitivity to radiographic contrast agents.
3. Subject with a pre-existing neurological or psychiatric disease that would confound the neurological and functional evaluations. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of hemorrhage on presentation.
4. CT or MRI ASPECT score of ≤6 in the anterior circulation, or pc-ASPECTS of ≤7.
5. CT or MRI evidence of mass effect or intra-cranial tumor (except small meningioma).
6. Current participation in another investigation drug or device treatment study.
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency.
8. Warfarin therapy with INR greater than 1.7.
9. Low molecular Weight Heparins, Heparin, Factor Xa inhibitors or direct thrombin inhibitors as full dose within the last 48 hours from screening and must have a normal partial thromboplastin time (PTT) to be eligible.
10. Baseline lab values: glucose < 50 mg/dL or > 400 mg/dL, platelets < 100,000 or Hct < 25.
11. Renal Failure as defined by a serum creatinine > 2.0 or Glomerular Filtration Rate [GFR]< 30.
12. Life expectancy of less than 90 days.
13. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal.
14. Presumed septic embolus, or suspicion of bacterial endocarditis.
15. Preprocedural or intraprocedural diagnosis of an unexpected vascular lesion or condition that may require additional, non-standard thrombectomy endovascular procedure(s), such as stenting, angioplasty or other treatment, and pose an additional or elevated risk. Such conditions, listed below, exclude or invalidate enrollment in the study:

    1. Previous intracranial hemorrhage, neoplasm, subarachnoid hemorrhage, cerebral aneurysm, or arteriovenous malformation
    2. Previously unknown dissection, vasculitis, vasculopathy, severe hemodynamically significant vascular stenosis, or other atypical vascular lesion
    3. Tandem lesions, defined as an occlusion involving both the cervical and intracranial segment of the same vascular distribution
    4. Stroke or vascular occlusions in multiple vascular territories

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females between 18-85 that present with acute ischemic strokes with large vessel occlusions and NIHSS<6.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic cerebral hemorrhage (ECASS definition) | Within 24 hours of intervention
  European Cooperative Acute Stroke Study (ECASS) classification: hemorrhagic infarct type 1 (HI1): small petechiae along the periphery of the infarct; hemorrhagic infarct type 2 (HI2): confluent petechiae within the infarcted area without a space-occupying effect; parenchymal hematoma type 1 (PH1): bleeding </= 30% of the infarcted area with a mild space-occupying effect. parenchymal hematoma type 2 (PH2): bleeding > 30% of the infarcted area with a significant space-occupying effect
Number of patients with a change in NIHSS by ≥ 4 points compared to enrollment NIHSS | Within 72 hours of intervention, or during hospitalization
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.

SECONDARY OUTCOMES:
Rate of successful angiographic recanalization grade TICI 2B or TICI 3 in the interventional arm | On the day of index procedure (Day 0). This will be assessed on the last angiographic run that is performed during the index intervention for the patient's stroke
  Thrombolysis in Cerebral Infarction (TICI) score: measures brain perfusion. Range 0-3. 0=no perfusion; 1= penetration, but no distal branch vessel filling; 2a= perfusion with incomplete (<50%) distal branch vessel filling; 2b=perfusion with incomplete (>50%) distal branch filling; 2c=perfusion with almost complete (>90%) distal branch filling; 3=full perfusion with filling of all distal branches
Global disability assessment via modified Rankin Score (mRS) in all patients | On the 1 day of discharge from hospitalization for the initial stroke event.
  Modified Rankin Score (mRS):a disability score with a range of 0-6. 0 = The patient has no residual symptoms. 1 = The patient has no significant disability, able to carry out all pre-stroke activities. 2 = The patient has slight disability, unable to carry out all pre-stroke activities but able to look after self without daily help. 3 = The patient has moderate disability, requiring some external help but able to walk without the assistance of another individual. 4 = The patient has moderately severe disability, unable to walk or attend to bodily functions without assistance of another individual. 5 = The patient has severe disability; bedridden, incontinent, requires continuous care. 6 = The patient has expired.
Final infarct volume on CT or MRI, change of infarct volume on CT or MRI, and CTA collateral scores | Repeat imaging within 2-5 days after event
  Volume measurement on imaging studies in milliliters (mm) or cubic centimeters (cm3)
Residual stroke symptom severity assessment via National Health Institute Stroke Scale (NIHSS) in all patients | On the 1 day of discharge from hospitalization for the initial stroke event.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Global disability assessment via modified Rankin Score (mRS) in all patients | 30 days after procedure
  Modified Rankin Score (mRS):a disability score with a range of 0-6. 0 = The patient has no residual symptoms. 1 = The patient has no significant disability, able to carry out all pre-stroke activities. 2 = The patient has slight disability, unable to carry out all pre-stroke activities but able to look after self without daily help. 3 = The patient has moderate disability, requiring some external help but able to walk without the assistance of another individual. 4 = The patient has moderately severe disability, unable to walk or attend to bodily functions without assistance of another individual. 5 = The patient has severe disability; bedridden, incontinent, requires continuous care. 6 = The patient has expired.
Residual stroke symptom severity assessment via National Health Instsitute Stroke Scale (NIHSS) in all patients | 30 days after procedure
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Toth, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share data.